CLINICAL TRIAL: NCT03775941
Title: Neuroprotective Effects of Cardiorespiratory Fitness on White Matter Integrity and Cognition Across the Adult Lifespan
Brief Title: Fitness on White Matter and Cognition in Aging
Status: Completed | Type: Observational
Sponsor: Suffolk University (Other)
Responsible Party: Principal Investigator, Ryan Mace, Clinical Psychology Doctoral Candidate, Suffolk University
Other Study IDs: NKI-RS; R01MH094639-01 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2018-12-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cognitive Decline; Executive Dysfunction; Cardiovascular Risk Factor
Keywords: Neuroimaging; White matter; Cardiorespiratory fitness; Physical activity; Cognitive aging; Executive function; Cognitive reserve
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-Sectional Lifespan Connectomics Study

SUMMARY:
Cardiorespiratory fitness (CRF) is associated with decreased risk for mild cognitive impairment (MCI) and dementia. CRF is linked with more conserved gray and white matter (WM) volume, improved WM microstructural integrity, and better cognitive performance among healthy older adults. Additional research is needed to determine: (1) which WM tracts are most strongly related to CRF, (2) whether CRF-related benefits on WM translate to enhanced cognitive functioning, and (3) factors that mediate and moderate CRF effects. Higher CRF was hypothesized to be associated with stronger WM integrity, both globally and locally in WM tracts that connect frontal brain regions. The neuroprotective effects were hypothesized to be age-dependent, such that the association between CRF and WM integrity would be stronger in old age compared to younger age. Finally, higher CRF was hypothesized to predict stronger performance on tests of executive functioning (EF), partially mediated by frontal WM integrity. Delineation of specific neurocognitive effects of CRF may serve clinicians in individually tailoring wellness interventions to meet patients' specific cognitive concerns with aging.

DETAILED DESCRIPTION:
Sample: Participant data from the "Cross-Sectional Lifespan Connectomics Study" of the Nathan Kline Institute - Rockland Sample (NKI-RS) will be analyzed for the present study. Zip code-based recruitment and monitoring enrollment for key demographic variables (e.g., age, sex, ethnicity) were used to maintain adequate representation of Rockland County and prevent sampling biases (e.g., cohort effects). NKI-RS eligibility was designed for inclusivity.

Procedure: All participants completed a medical evaluation, psychiatric interview, self-report questionnaires, standardized battery of cognitive tests, and neuroimaging at NKI. Complete details about the MRI measurement parameters can be located on the NKI-RS website for DTI and MPRAGE and protocols. Quality assurance of raw data, inclusive of monitoring standard operating procedures, error-handling, and compiling the data dictionary, is maintained by NKI-RS. Raw neuroimaging data was acquired by NKI-RS and processed at Suffolk University using TRACULA and FreeSurfer 5.3.

Statistical Plan: Analyses will be performed on de-identified phenotypic and neuroimaging data from adult NKI-RS participants available at the start of this study (October 2016). Analyses will evaluate the potential for CRF to modulate decline in WM integrity and EF observed with aging. Mixed-effects modeling will investigate the extent to which CRF predicts WM integrity, as both a global measurement of fractional anisotropy (FA) and FA within nine major WM tracts. Structural equation modeling will examine whether higher FA within frontal WM tracts partially mediates a positive relationship between CRF and EF. The role of age and clinical characteristics (e.g., cardiovascular risk factors, depression) will also be explored as covariates in the link between CRF, WM, and EF.

ELIGIBILITY:
NKI-RS eligibility criteria was designed for inclusivity. Nearly half of recruited individuals met criteria for at least one Diagnostic Statistical Manual - 4th Edition diagnosis based on a semi-structured clinical interview.

Inclusion Criteria (present study):

* diffusion tensor imaging (DTI) without significant artifacts
* T1-weighted structural imaging (Magnetization-Prepared Rapid Gradient-Echo; MPRAGE) without significant artifacts
* CRF data from a standardized cycle ergometer test (commonly used for predicting maximal oxygen uptake; VO2 max).

Exclusion Criteria (per NKI-RS protocol):

* severe psychiatric illness (bipolar disorder, schizophrenia disorder, schizoaffective disorder)
* severe developmental disorders (autism spectrum disorders, intellectual disabilities)
* current suicidal or homicidal ideation
* severe cerebral trauma (stroke, moderate to severe traumatic brain injury, ischemic attack in the past two years)
* severe neurodegenerative disorders (Parkinson's disease, Huntington's Disease, dementia)
* a history of substance dependence in the past two years (with an exception for cannabis)
* a lifetime history of psychiatric hospitalization
* current pregnancy
* MRI contraindications

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are community-dwelling adults from the "Cross-Sectional Lifespan Connectomics Study" of the Nathan Kline Institute - Rockland Sample (NKI-RS)-a large cross-sectional sample of adult brain development. NKI prospectively recruited community-dwelling residents of Rockland County, New York-a region that is socioeconomically comparable to United States demographics.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07

PRIMARY OUTCOMES:
white matter (WM) microstructure integrity | Measured between 9:00 and 10:00 am on the single assessment day.
  fractional anisotropy (FA) diffusion tensor imaging (DTI)
executive function (EF) | Measured between 12:30 and 2:30 pm on the single assessment day.
  Delis-Kaplan Executive Function System (D-KEFS) subtests will include the Trail Making Test, Design Fluency Test, Color-Word Interference Test, and Tower Tests. Scores from each subtest will be transformed into z-scores to yield the same units of measurement. Then, structural equation modeling (SEM) will aggregate these values quantify a construct of overall EF.
executive function (EF) | Measured between 11:00 am and 12:00 pm on the single assessment day.
  Penn Computerized Neurocognitive Battery (CNB) subtests will include the CNB Letter N-back Test and Conditional Exclusion Test. Scores from each subtest will be transformed into z-scores to yield the same units of measurement. Then, structural equation modeling (SEM) will aggregate these values quantify a construct of overall EF.

IPD SHARING:
Plan to Share IPD: Yes
The Nathan Kline Institute - Rockland Sample is a public, open-access data repository that is available upon approval of the NKI data usage agreement.
  R code for all study analyses will be made available for reproducibility with open-access NKI-RS data.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Nooner KB, Colcombe SJ, Tobe RH, Mennes M, Benedict MM, Moreno AL, Panek LJ, Brown S, Zavitz ST, Li Q, Sikka S, Gutman D, Bangaru S, Schlachter RT, Kamiel SM, Anwar AR, Hinz CM, Kaplan MS, Rachlin AB, Adelsberg S, Cheung B, Khanuja R, Yan C, Craddock CC, Calhoun V, Courtney W, King M, Wood D, Cox CL, Kelly AM, Di Martino A, Petkova E, Reiss PT, Duan N, Thomsen D, Biswal B, Coffey B, Hoptman MJ, Javitt DC, Pomara N, Sidtis JJ, Koplewicz HS, Castellanos FX, Leventhal BL, Milham MP. The NKI-Rockland Sample: A Model for Accelerating the Pace of Discovery Science in Psychiatry. Front Neurosci. 2012 Oct 16;6:152. doi: 10.3389/fnins.2012.00152. eCollection 2012. PMID 23087608
- [Derived] Andrade MA, Raposo A, Andrade A. Exploring the late maturation of an intrinsic episodic memory network: A resting-state fMRI study. Dev Cogn Neurosci. 2024 Dec;70:101453. doi: 10.1016/j.dcn.2024.101453. Epub 2024 Sep 26. PMID 39368283
- See also: US Census Bureau. (2010). U.S. Census Bureau State & County Quickfacts. — https://www.census.gov/quickfacts/
- See also: NKI-RS DTI protocol — http://fcon_1000.projects.nitrc.org/indi/pro/eNKI_RS_TRT/DIff_137.pdf
- See also: NKI-RS MPRAGE protocol — http://fcon_1000.projects.nitrc.org/indi/enhanced/NKI_MPRAGE.pdf
- See also: NKI-RS data usage agreement — http://fcon_1000.projects.nitrc.org/indi/enhanced/access.html